CLINICAL TRIAL: NCT04711707
Title: Addressing the Social Needs of Children Attending a Weight Management Program: a Pilot Randomized Controlled Trial
Brief Title: Addressing the Social Needs of Children With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 12697
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obesity, Childhood
Keywords: Social Determinants of Health; Obesity; Child Health; Social needs
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Participants who screen positive for social needs will be randomized to receive one of two possible interventions. An allocation ratio of 1:1 with random permuted blocks of varying size will be used. Random block size will help to ensure that investigators or outcome assessors will not be able to decipher the block size and anticipate future allocations. Allocation concealment is the process that prevents any trial participant or investigator from knowing in advance the treatment to which subjects will be assigned and seeks to prevent selection bias.
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blind to the group allocation. Group allocation will be concealed until the final data analysis is performed. Families, research staff and clinical staff will not be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community navigator (Experimental): This group is guided through the resources and provided bi-monthly support with a community navigator
  Interventions: Other: Community navigator
- Self-Navigation (Other): This group receives the social needs resources to self-navigation
  Interventions: Other: Self-Navigation

INTERVENTIONS:
Other: Community navigator — All patients who consent to participate in the study will complete a pediatric social history tool to identify social needs. The intervention group will receive support through a community navigator to guide and understand appropriate services for their specific needs. This arm will receive guidance and bimonthly check-ins.
  Arms: Community navigator
Other: Self-Navigation — The control group will receive an electronic or paper copy of community resources that address the identified social needs.
  Arms: Self-Navigation

SUMMARY:
This study aims to improve the treatment of a common, chronic health concern for children: obesity. It has the potential to improve the care we provide by testing an intervention that addresses social needs and the important upstream factors that influences health outcomes.

DETAILED DESCRIPTION:
Addressing the social needs of children attending a weight management program. The specific aims of this pilot randomized controlled trial are the following:

1. To determine the feasibility of implementation and delivery of a screening-referral intervention versus usual care to address social needs of children with obesity enrolled in a pediatric weight management program at McMaster Children's Hospital, which will include recruitment rates, uptake of the intervention, and follow-up of participants.
2. To understand impact on health outcomes of a screening-referral intervention versus usual care to address social needs of children with obesity enrolled in a pediatric weight management program including change in i) body mass index z score (zBMI); ii) change in body composition; and iii) change in health-related quality of life.

Hypothesis: We hypothesize that health outcomes of children with obesity are connected to the social determinants of health, and that an intervention which screens for and refers to community supports will improve child obesity outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the weight management program

Exclusion Criteria:

* Children in the care of child protection services and/or living in group or foster care. Children in these settings will not be living within typical family-systems to have social needs addressed by this intervention.
* Parents who cannot read and write in English

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | 6 months
  Recruitment rate refers to the number of participants enrolled and is measured by the number of consent forms signed or implied. Recruitment will be successful if 80% of our target sample is met.
Uptake of Intervention | 6 months
  Uptake of the intervention refers to the number of enrolled families who completed all aspect of the intervention. Elements that are part of the uptake include: social history following enrollment as well as the quality of life questionnaires and use of service questionnaire at enrolment and 6-months. Uptake will be considered successful if >80% of families complete the intervention.
Follow-up of Participants | 6 months
  Follow-up of participants refers to the participants attending all of their scheduled study visits. The study will be considered successful if >90% of participants complete all study visits.

SECONDARY OUTCOMES:
Change in Body Mass Index Z-Score | 6 Months
  The body mass index Z-score (zBMI) is calculated using WHO growth charts, for age and sex. Height and weight of the child will be collected from the chart at baseline and from every visit the participant has in clinic until the end of the intervention. BMI will be calculated by dividing weight in kilograms by the square of the body height in metres squared.
Change in Body Composition | 6 Months
  Body fat will be assessed at baseline and at the end of the intervention using the Quantum II BIA analyzer (RJL Systems). Bioelectrical impedance analysis (BIA) is non-invasive and portable. It measures electrical impedance of tissues by applying alternating current to the body tissues (not felt by the participant), which is used in regression equations to approximate body fat and fat free mass. This will be collected at baseline from the chart and from every visit the participant has in clinic until the end of the intervention.
Change in Quality of Life | 6 Months
  Quality of life will be measured using the Pediatrics Quality of Life Inventory (PedsQL™). Both the patient and the parent or guardian will be asked to complete the PedsQL™. The minimum possible score for this inventory is 0 and the highest is 100. Higher scores indicate a better Health Related Quality of Life (HRQOL).

CONTACTS AND LOCATIONS:
Overall Officials: Gita Wahi, MD, MSc, Principal Investigator — McMaster Children's Hospital
Locations (1):
- Kimberley Krasevich, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The data collected for the purposes of this study will only be made available to the principal investigator, co-investigators and the research staff associated with the study.

REFERENCES:
- [Background] Oliver LN, Hayes MV. Neighbourhood socio-economic status and the prevalence of overweight Canadian children and youth. Can J Public Health. 2005 Nov-Dec;96(6):415-20. doi: 10.1007/BF03405180. PMID 16350864
- [Background] Hadjiyannakis S, Ibrahim Q, Li J, Ball GDC, Buchholz A, Hamilton JK, Zenlea I, Ho J, Legault L, Laberge AM, Thabane L, Tremblay M, Morrison KM. Obesity class versus the Edmonton Obesity Staging System for Pediatrics to define health risk in childhood obesity: results from the CANPWR cross-sectional study. Lancet Child Adolesc Health. 2019 Jun;3(6):398-407. doi: 10.1016/S2352-4642(19)30056-2. Epub 2019 Apr 3. PMID 30952624
- [Background] COUNCIL ON COMMUNITY PEDIATRICS. Poverty and Child Health in the United States. Pediatrics. 2016 Apr;137(4):e20160339. doi: 10.1542/peds.2016-0339. Epub 2016 Mar 9. PMID 26962238
- [Background] Gottlieb LM, Wing H, Adler NE. A Systematic Review of Interventions on Patients' Social and Economic Needs. Am J Prev Med. 2017 Nov;53(5):719-729. doi: 10.1016/j.amepre.2017.05.011. Epub 2017 Jul 5. PMID 28688725
- [Background] Fox CK, Cairns N, Sunni M, Turnberg GL, Gross AC. Addressing Food Insecurity in a Pediatric Weight Management Clinic: A Pilot Intervention. J Pediatr Health Care. 2016 Sep-Oct;30(5):e11-5. doi: 10.1016/j.pedhc.2016.05.003. Epub 2016 Jun 16. PMID 27321679
- [Background] Fazalullasha F, Taras J, Morinis J, Levin L, Karmali K, Neilson B, Muskat B, Bloch G, Chan K, McDonald M, Makin S, Ford-Jones EL. From office tools to community supports: The need for infrastructure to address the social determinants of health in paediatric practice. Paediatr Child Health. 2014 Apr;19(4):195-9. doi: 10.1093/pch/19.4.195. PMID 24855416
- [Background] Kenyon C, Sandel M, Silverstein M, Shakir A, Zuckerman B. Revisiting the social history for child health. Pediatrics. 2007 Sep;120(3):e734-8. doi: 10.1542/peds.2006-2495. No abstract available. PMID 17766513
- [Background] Colvin JD, Bettenhausen JL, Anderson-Carpenter KD, Collie-Akers V, Plencner L, Krager M, Nelson B, Donnelly S, Simmons J, Higinio V, Chung PJ. Multiple Behavior Change Intervention to Improve Detection of Unmet Social Needs and Resulting Resource Referrals. Acad Pediatr. 2016 Mar;16(2):168-74. doi: 10.1016/j.acap.2015.06.001. Epub 2015 Jul 14. PMID 26183003
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Chen E, Martin AD, Matthews KA. Trajectories of socioeconomic status across children's lifetime predict health. Pediatrics. 2007 Aug;120(2):e297-303. doi: 10.1542/peds.2006-3098. Epub 2007 Jul 2. PMID 17606533
- [Background] Ligthart KAM, Buitendijk L, Koes BW, van Middelkoop M. The association between ethnicity, socioeconomic status and compliance to pediatric weight-management interventions - A systematic review. Obes Res Clin Pract. 2017 Sep-Oct;11(5 Suppl 1):1-51. doi: 10.1016/j.orcp.2016.04.001. Epub 2016 Apr 20. PMID 27108215
- [Derived] Wahi G, Marjerrison S, Gill S, Krasevich K, Morrison KM, Thabane L. Addressing unmet social needs of children with obesity: a pilot randomized controlled trial. Pilot Feasibility Stud. 2024 Nov 14;10(1):141. doi: 10.1186/s40814-024-01570-9. PMID 39543718
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077
- [Derived] Wahi G, Marjerrison S, Gutierrez C, Krasevich K, Morrison KM, Thabane L. Screening and addressing social needs of children and families enrolled in a pediatric weight management program: a protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Jun 18;8(1):129. doi: 10.1186/s40814-022-01080-6. PMID 35717284
- See also: The World Health Organization's Department of Social Determinants of Health webpage. It provides information about the social, physical and economic conditions in society that impact upon health. — http://www.who.int/social_determinants/sdh_definition/en/
- See also: Produced by Public Health Ontario, tt provides access to the Ontario Marginalization Index (ON-MARG). ON-MARG is a multifaceted index which measures axes of deprivation in Ontario, including economic, ethno-racial, age based and social. — http://www.publichealthontario.ca/en/data-and-analysis/health-equity/ontario-marginalization-index
- See also: Access to an electronic database of Ontario's government and community based social services. — http://211ontario.ca/